CLINICAL TRIAL: NCT03287856
Title: Investigation of the Safety and Performance of the NVT ALLEGRA TAVI System TF in Patients With Failed Surgical Aortic Bioprosthesis and Elevated Surgical Risk
Brief Title: NVT ALLEGRA TAVI System TF in Failing Surgical Aortic Bioprosthesis
Acronym: VIVALL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NVT GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NVT03VIV
Record Dates: First submitted 2017-08-15; First posted 2017-09-19 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Transcatheter Aortic Valve Implantation
Keywords: Valve-in-valve; TAVI
MeSH Terms: interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Transcatheter Aortic Valve Implantation (TAVI) in failing surgical bioprosthesis
  Interventions: Device: Transcatheter Aortic Valve Implantation (TAVI)

INTERVENTIONS:
Device: Transcatheter Aortic Valve Implantation (TAVI) — Implantation of the ALLEGRA Transcatheter Heart Valve in failing surgical bioprosthesis

SUMMARY:
The study investigates the technical feasibility of the replacement of failed surgical bioprosthetic aortic valves by the ALLEGRA Transcatheter Heart Valve (THV) and describes the safety and performance profile

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* Symptomatic degeneration of aortic bioprosthesis showing echocardiographically mean aortic gradient >40mmHg or peak jet velocity >4.0m/s and AVA<1.0cm2 OR symptomatic patients with severe bioprosthetic valve insufficiency.
* High risk for redo surgery defined by STS ≥10% / EuroScore II ≥7% OR as assessed by the heart team
* Has signed the Patient Informed Consent Form
* Willing and able to comply with requirements of the study, including all follow-up visits
* Female patients of childbearing potential have a negative pregnancy test ≤7 days before the procedure and are willing to use a reliable method of birth control for the duration of study participation

Exclusion Criteria:

* Low position of the coronary ostia, especially in combination with shallow sinuses
* Echocardiographic evidence of intracardiac mass, thrombus or vegetation
* Significant aortic disease such as severe obstructive calcification or marked tortuosity or kinking which will preclude a safe advancement of the ALLEGRA TAVI System TF
* Iliofemoral vessel conditions such as severe obstructive calcification, severe tortuosity or kinking that would preclude safe placement of an 18 Fr introducer sheath or make endovascular access to the aortic valve impossible
* Severe mitral insufficiency
* Internal diameter of the bioprosthesis is ≤16 mm or >28 mm
* Patient prosthesis mismatch (EOAi ≤0.65 cm2/m2) as the underlying cause of the poor valve function and need for re-intervention
* Non-valvular stenosis as the underlying cause of the poor valve function and need for re-intervention
* Failing pre-existing prosthetic heart valve or prosthetic ring in any other position than aortic
* Partially detached leaflets that in the aortic position may obstruct a coronary ostium.
* Existence of aortic conduit, aortic arch replacement, stentless bioprosthesis and autologous valve replacement
* Paravalvular leak of the failing surgical bioprosthesis (between failing surgical bioprosthesis and native annulus)
* LVEF <20%
* Evidence of active endocarditis or other acute infections
* End stage renal disease requiring chronic dialysis or creatinine clearance <20 ml/min or serum creatinine >3.0 mg/dl (264 µmol/l)
* Known hypersensitivity to contrast media, which cannot be adequately pre-medicated or contraindication to anticoagulant or anti-platelet medication or to Nitinol alloy or to bovine tissue
* Evidence of an acute myocardial infarction within the past 30 days
* Cerebral vascular accident (TIA, Stroke) within past 6 months (≤180 days)
* Evidence of active peptic ulcer or upper gastrointestinal bleeding within past 90 days
* Untreated clinically significant coronary artery disease requiring revascularization
* Hemodynamic instability (e.g. cardiogenic shock) requiring inotropic support or mechanical heart assistance (e.g. VAD, IABP)
* Uncontrolled (therapy resistant) atrial fibrillation
* Need for emergency surgery for any reason
* Life expectancy ≤ 12 months due to other medical illness
* Currently participating in another investigational drug or device study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-11 (Actual); Primary Completion 2018-09-27 (Actual); Study Completion 2019-10-27 (Actual)

PRIMARY OUTCOMES:
Mean pressure gradient | immediately after index-procedure
30-days survival | 30 days
  Proportion of participants with overall survival at 30 days

SECONDARY OUTCOMES:
Cardiovascular mortality | 30 days
Hemodynamic parameters | up to12 months
  pressure gradient, effective orifice area, velocity
Technical success of implantation | immediately after index-procedure
  defined as absence of procedural mortality AND correct positioning of a single prosthetic heart valve into the proper anatomical location AND no severe (<0.65 cm2/m2) prosthesis - patient mismatch AND mean aortic valve gradient <20 mmHg AND no moderate or severe prosthetic valve regurgitation
Early safety | 30 days
  all-cause mortality, all stroke (disabling and non-disabling), life-threatening bleeding, acute kidney injury stage 2 or 3 (including renal replacement therapy), coronary artery obstruction requiring Intervention, major vascular complication, valve-related dysfunction requiring repeat procedure
Time related valve safety | up to 12 months
  structural valve deterioration as defined by
  * requiring repeat procedure (transcatheter or surgical heart valve replacement)
  * valve-related dysfunction defined by
    * mean aortic valve gradient ≥20 mmHg AND
    * no moderate or severe prosthetic valve regurgitation
New Pacemaker implantation | up to 12 months
  Proportion of patients with pacemaker implantations after index-procedure
NYHA classification | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Schaefer, MD, Principal Investigator — Universitäres Herzzentrum Hamburg, Germany
Locations (5):
- Germany (5):
  - Segeberger Kliniken, Herzzentrum, Bad Segeberg
  - Immanuel Klinik Bernau Herzzentrum Brandenburg, Bernau bei Berlin
  - Mitteldeutsches Herzzentrum Universitätsklinikum Halle (Saale), Halle
  - Asklepios Klinik St. Georg, Hamburg
  - Universitäres Herzzentrum Hamburg GmbH, Hamburg

REFERENCES:
- [Result] Schafer U, Butter C, Landt M, Frerker C, Treede H, Schirmer J, Koban C, Allali A, Schmidt T, Charitos E, Conradi L. Thirty-day outcomes of a novel transcatheter heart valve to treat degenerated surgical valves: the VIVALL multicentre, single-arm, pilot study. EuroIntervention. 2019 Oct 4;15(9):e757-e763. doi: 10.4244/EIJ-D-19-00331. PMID 31355750
- See also: Related Info — https://eurointervention.pcronline.com/article/thirty-day-outcomes-of-a-novel-transcatheter-heart-valve-to-treat-degenerated-surgical-valves-the-vivall-multi-center-single-arm-pilot-study